CLINICAL TRIAL: NCT03754634
Title: A Prospective, Open, Multicenter Clinical Trial of Eltrombopag Combined With Diacerein in the Management of Eltrombopag-inefficient or Relapsed ITP
Brief Title: A Prospective, Open, Multicenter Clinical Trial of Eltrombopag Combined With Diacerein in Eltrombopag-inefficient or Relapsed ITP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other); Anhui Medical University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shenzhen Second People's Hospital (Other); Zhejiang Provincial Hospital of TCM (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Diacerein
Record Dates: First submitted 2018-11-25; First posted 2018-11-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Thrombocytopenia
Keywords: ITP; Eltrombopag; Diacerein
MeSH Terms: conditions — Thrombocytopenia | interventions — eltrombopag; diacerein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- drugs (Experimental): Eltrombopag and Diacerein
  Interventions: Drug: Eltrombopag and Diacerein

INTERVENTIONS:
Drug: Eltrombopag and Diacerein — The initial dose of eltrombopag administration is 25 mg orally once daily, which could be transited to 50 mg/d in a 2-week cycle according to the need, and the maximum dose was not more than 75 mg/d. The dose of diacerein administration is 50 mg orally twice daily. The treatment was discontinued after 6 weeks without blood index reaction.
  Other Names: diacetylrhein

SUMMARY:
Eltrombopag is an oral thrombopoietin receptor agonist that has been licensed for use as second line therapy in ITP patients. Diacerein is a slow-acting medicine of the class anthraquinone used to treat joint diseases such as osteoarthritis. The project was undertaking by Qilu Hospital of Shandong University and other 5 well-known hospitals in China. In order to report the efficacy and safety of eltrombopag combined with diacerein in the management of ITP.

DETAILED DESCRIPTION:
The investigators are undertaking a prospective, open, multicentre trial of 30 ITP adult patients with eltrombopag-inefficient or relapsed from 6 medical centers in China. The initial dose of eltrombopag administration is 25 mg orally once daily, which could be transited to 50 mg/d in a 2-week cycle according to the need, and the maximum dose was not more than 75 mg/d. The dose of diacerein administration is 50 mg orally twice daily. The treatment was discontinued after 6 weeks without blood index reaction.

Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. In order to report the efficacy and safety of eltrombopag combined with diacerein for the treatment of adults patients with eltrombopag-inefficient or relapsed.

ELIGIBILITY:
Inclusion Criteria:

* ITP patients with eltrombopag-inefficient or relapsed need of treatment(s) to minimize the risk of clinically significant bleeding primary ITP confirmed by excluding other supervened causes of thrombocytopenia

Exclusion Criteria:

* pregnancy hypertension cardiovascular disease diabetes liver and kidney function impairment HCV, HIV, HBsAg seropositive status patients with systemic lupus erythematosus and/or antiphospholipid syndrome

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of platelet response | the sixth weeks
  R. A response (R) was defined as platelet count ≥ 30×10^9/L without bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Result] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Result] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182